CLINICAL TRIAL: NCT06291259
Title: Mpox Prospective Observational Cohort Study
Acronym: MPOCS
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: CTO 4081
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Monkeypox
Keywords: mpox
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Acute phase:
  1. Blood
  2. Urine
  3. Nasopharyngeal swab
  4. Throat swab
  5. Rectal swab
  6. Semen sample or vaginal swab, as applicable
  7. Skin lesions (see below)
  8. Breastmilk, if lactating
  Convalescent phase:
  1. Rectal swab
  2. Semen sample/vaginal swab (as applicable)
  3. Breastmilk (if applicable).
  Samples are collected for testing of mpox PCR and serology.
  Participants will be asked to consent to storage of these samples for future testing as well (e.g. biobanking)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Confirmed positive for mpox: Participants with laboratory test results confirming the diagnosis of Mpox. This includes the total number of unique participants who complete the main part 1 study, those who complete the baseline visit only, those who agree to frequent sampling, and those who only participate in part 2.
- Confirmed negative for mpox: Participants in whom the clinician feels that the diagnosis of Mpox has been clearly ruled out.

SUMMARY:
The goal of this multicentre prospective observational cohort study is to shed light on the following unknowns:

1. The clinical manifestations of Mpox infection since the 2022 outbreak in Canada.
2. The social and psychological impacts of Mpox infection since the 2022 outbreak in Canada
3. The transmissibility of Mpox infection
4. Viral shedding over time in infected individuals

The study is divided into Part 1 (corresponding to the acute phase of illness) and Part 2 (corresponding to the convalescent phase of the illness); part 2 will be optional. Participants enrolled during the acute phase of illness will complete part 1 of the study and will be invited to participate in Part 2 as well. Part 1 of the study will include the following three core components, at baseline and weekly (±3 days) until one week after the resolution of all symptoms (i.e. one week after complete healing of skin lesions):

1. Collection of clinical data through chart review and research staff interviews with study participants
2. Participant self-administered online questionnaires at baseline and a thrice-weekly 'acute phase participant diary'
3. Specimen collection for Mpox-related testing Optional components for Part 1 include baseline-only, questionnaire-only, and frequent sampling.

Other optional components for all participants include in the Image Atlas, an online database of clinical images of mpox, designed to provide clinicians and community members of what mpox looks like in real life, and the biobank, which will store research samples for potential future studies.

DETAILED DESCRIPTION:
Mpox is caused by a virus that normally infects animals (rodents, monkeys, and others), but can sometimes infect humans. In the past, it was usually only seen in a few specific countries, but since the beginning of May 2022 it has been reported in many other countries, including Canada, where it has never been seen before. The virus can cause several symptoms, including "flu-like" symptoms (fever, headache, feeling tired, muscle pains, swollen glands, sore throat) and skin symptoms (spots, bumps, blisters, open sores, scabs). However, sometimes it can also cause very few symptoms, or no symptoms at all. Mpox can be spread from one person to another in a few ways, such as directly touching the affected skin areas of someone who has the infection, touching sheets or clothes that were used by someone with the infection, or breathing in particles of virus that came from the nose, mouth and lungs of someone with the infection ("respiratory droplets").

In the cases seen around the world since May 2022, doctors and patients have noticed many things that are unusual for mpox infection. Some of these relate to the symptoms people have had (for example, the order in which people get different symptoms might be changing), and the ways in which it has been spread from person to person (for example, we do not know if it can be spread through sex). There is also worry that the infection could have bad effects on people's financial situation and emotional wellness, especially because people with mpox have to self-isolate at home for several days or weeks until the infection is completely over, to protect public health. Finally, there is also a lot that doctors and scientists still do not yet know about the virus itself, including the specific parts of the body where it can be found, the amount of time that it stays in those parts of the body, and its biology (e.g. its "genetic sequence" or genes).

The purpose of this study is to learn more about 1) the symptoms people have, 2) the ways mpox is spread, 3) the effects on people's lives, and 4) the virus itself, including the places in the body and surrounding environment where it can live. Canada is currently experiencing an outbreak and the outlined purposes are critical and relevant to clinical and public health control efforts.

The study is divided into Part 1 (corresponding to the acute phase of illness) and Part 2 (corresponding to the convalescent phase of the illness); part 2 will be optional. Participants enrolled during the acute phase of illness will complete part 1 of the study and will be invited to participate in Part 2 as well. Part 1 of the study will include the following three core components, at baseline and weekly (±3 days) until one week after the resolution of all symptoms (i.e. one week after complete healing of skin lesions):

1. Collection of clinical data through chart review and research staff interviews with study participants
2. Participant self-administered online questionnaires at baseline and a thrice-weekly 'acute phase participant diary'
3. Specimen collection for Mpox-related testing Optional components for Part 1 include baseline-only, questionnaire-only, and frequent sampling.

Other optional components for all participants include in the Image Atlas, an online database of clinical images of mpox, designed to provide clinicians and community members of what mpox looks like in real life, and the biobank, which will store research samples for potential future studies.

ELIGIBILITY:
Inclusion Criteria

Part 1:

• Being investigated for Mpox infection by a clinician based on clinical (i.e. symptoms) and/or epidemiologic (i.e. exposure to confirmed case) grounds;

Part 2:

* Clinically confirmed to be in the convalescent phase (i.e. confirmed for Mpox infection previously)
* Within 12 weeks of symptom onset

Exclusion Criteria

• None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our overarching goal is to characterize key clinical and epidemiologic aspects of Mpox infection in Canada in the context of the rapidly emerging outbreak. As such we will deliberately include people both with (n=250) and without (number to be determined based on accrual of confirmed cases) the condition of interest because it is important to have a comparison group of people who are ultimately confirmed not to have the infection
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Description of clinical manifestation | 12 weeks
  Clinical manifestations of mpox infection during the Canadian outbreak, including symptom duration and spectrum, complications, natural history and sources of variability in clinical manifestations
Psychosocial impact | 12 weeks
  Describe the psychosocial impacts of mpox-related illness and isolation requirements, including financial insecurity, psychological distress and perceived and enacted stigma
Transmission-related aspects of mpox infection | 12 weeks
  Types and timing of human and animal contacts prior to mpox infection, as well as quantifying the detectability of mpox viral DNA in the immediate environment of people ultimately diagnosed with the infection, including physical surfaces and air samples
Virologic aspects of mpox infection over time | 12 weeks
  Detectability of mpox viral DNA by polymerase chain reaction (PCR) along with the associated cycle threshold, as well as titers of infectious virus, in different anatomic compartments and examining the viral genomic sequence. Outcomes also include characterizing the host response to mpox infection including host gene and cytokine expression and antibody titers.

CONTACTS AND LOCATIONS:
Overall Officials: Darrell HS Tan, MD, Principal Investigator — Unity Health Toronto
Locations (3):
- Canada (3):
  - BC Centre For Excellence, Vancouver, British Columbia
  - Unity Health Toronto, Toronto, Ontario
  - University Health Network, Toronto, Ontario